CLINICAL TRIAL: NCT04960605
Title: Prognosis of Dental Implants in Patients With Primary Sjögren's Syndrome. A Prospective Study
Brief Title: Prognosis of Dental Implants in Patients With Primary Sjögren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: ITI Foundation (Industry); Gigtforeningen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mandana Hosseini, Guest researcher, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1036_2015
Record Dates: First submitted 2021-06-14; First posted 2021-07-14 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Dental Implant; Primary Sjögren Syndrome
Keywords: Dental Implants; Primary Sjögren syndrom; Biological outcome; Technical outcome; Aesthetic outcome; Patient-reported outcome
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: Prospective study
Who Masked: Outcomes Assessor
Masking Description: The statistical analyses will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Other): Patients with Primary Sjögren Syndrom
  Interventions: Procedure: Dental implants
- Control group (Other): Patients with Primary Sjögren Syndrom, matched to the test group
  Interventions: Procedure: Dental implants

INTERVENTIONS:
Procedure: Dental implants — Treatment of the toothless regions with dental implants

SUMMARY:
Primary Sjögren's Syndrome (PSS) is a chronic autoimmune inflammatory disease primarily involving the salivary and lacrimal glands. Few data exist regarding survival and success rate of dental implants in patients with PSS. Although a previous study suggest lower success rate for dental implants we hypothesize that dental implants have similar survival and success rate in PSS as healthy controls.

The purpose of the present study was to evaluate the long-term survival and success rate of dental implants in patients with PSS compared to the healthy controls.

DETAILED DESCRIPTION:
Sjögren's syndrome (SS) affects about 5% of population worldwide. Patients with Primary Sjögren's Syndrome (PSS) have dry mouth, oral mucosal problems, increased dental decay and problems wearing dentures. A retrospective case series indicated that implant survival rate may be reduced among SS patients. Furthermore, there is lack of scientific evidence to support success or failure of dental implants in SS-patients.

The null hypothesis is that the outcome of implant treatment after 5 years is similar in patients with primary Sjögren's Syndrome (pSS) compared to matched controls.

The participants with PSS fulfilled the Copenhagen Criteria and/or the US-EU criteria for PSS, miss at least one tooth and have sufficient bone volume for a single implant insertion without bone augmentation.

Recruitment of PSS patients was done via own existing databases on PSS patients as well as repeated national announcements in the Danish Dental Journal.

We included 24 consecutive participants with PSS. For each participant with PSS (test group), an age, gender, and tooth-type matched healthy participant (control group) was enrolled (n=24).

The surgical part of the implant treatment was carried out by two experienced maxillofacial surgeons. Straumann implants (Straumann Bone level Roxolid®) with a hydrophilic sandblasted, acid etched implant surface (SLActive) was used for all participants. If more than one implant was placed, the study implant was determined according to a randomization scheme.

The inserted implants were allowed to heal for 3 months before the prosthetic part, which was carried out by two experienced prostodontists. The same prosthetic material and method was applied for all participants.

The participants were recalled for baseline (2 months after prosthetic loading) and 1, 3 and 5 years examination, where the biological (marginal bone level, inflammation etc.), technical (fractures, loosening's etc.), esthetic (Copenhagen Index score) and patient-reported (Oral Health Impact Profile questionnaire/OHIP-49) assessments were performed.

ELIGIBILITY:
Inclusion Criteria:

* - Age 20-70 years
* Indication of tooth replacement with implant-supported fixed dentures
* The test group should be without any potentially associated disease
* pSS must be diagnosed according to the American-European Consensus Group criteria (Vitali et al., 2002):

  1. The presence of any 4 of the following 6 items, as long as either item IV (Histopathology) or VI (Serology) is positive
  2. The presence of any 3 of the 4 objective criteria items (that is, items III, IV, V, VI)

The items:

I. Ocular symptoms: a positive response to at least one of the following questions:

1. Have you had daily, persistent, troublesome dry eyes for more than 3 months?
2. Do you have a recurrent sensation of sand or gravel in the eyes?
3. Do you use tear substitutes more than 3 times a day?

II. Oral symptoms: a positive response to at least one of the following questions:

1. Have you had a daily feeling of dry mouth for more than 3 months?
2. Have you had recurrently or persistently swollen salivary glands as an adult?
3. Do you frequently drink liquids to aid in swallowing dry food?

III. Ocular signs --that is, objective evidence of ocular involvement defined as a positive result for at least one of the following two tests:

1. Schirmer's I test, performed without anaesthesia (<5 mm in 5 minutes)
2. Rose bengal score or other ocular dye score (>4 according to van Bijsterveld's scoring system) IV. Histopathology: In minor salivary glands (obtained through normal-appearing mucosa) focal lymphocytic sialoadenitis, evaluated by an expert histopathologist, with a focus score >1, defined as a number of lymphocytic foci (which are adjacent to normal-appearing mucous acini and contain more than 50 lymphocytes) per 4 mm2 of glandular tissue

V. Salivary gland involvement: objective evidence of salivary gland involvement defined by a positive result for at least one of the following diagnostic tests:

1. Unstimulated whole salivary flow (<1.5 ml in 15 minutes)
2. Parotid sialography showing the presence of diffuse sialectasias (punctate, cavitary or destructive pattern), without evidence of obstruction in the major ducts
3. Salivary scintigraphy showing delayed uptake, reduced concentration and/or delayed excretion of tracer

VI. Autoantibodies: presence in the serum of the following autoantibodies:

1. Antibodies to Ro(SSA) or La(SSB) antigens, or both

* The control group should match the test group according to the age, sex and treatment region and fulfill the following:
* Normal salivary flow: unstimulated > 1.5 ml in 15 min, stimulated > 3.5 ml in 5 min
* No ocular or oral symptoms
* Submission of written informed consent form

Exclusion Criteria:

* Persons with:

  1. secundary Sjögren Syndrom (sSS)
  2. severe systemic disease including severe bleeding disorder and/or conditions which put the patient at risk and/or prohibit compliance as stated by Hwang and Wang, 2006; and Hwang and Wang, 2007):
  3. previous or present bisphosphonate, Denosumab or anti-angiogenetic chemotherapeutic drugs
  4. poor bone quality according to Lekholm U & Zarb GA (1985) or diagnosed osteoporosis
  5. Heavy smokers, eqv. to 20+ cigarettes/day
  6. Noncompliance

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Number of patients with Sjögren syndrom | Five years
  number of participants in the test group
Number of patients without Sjögren syndrom | Five years
  number of participants in the control group
Number of implants in each group | Five years
  number of implants in patients with or without Sjögren syndrom
Marginal bone loss | Five years
  Marginal bone level change over the time in millimeter: radiological examinations and measurements of the marginal bone at implants mesially and distally (millimeter) and the change of the marginal bone level between different observation
Frequency of implant sites with biological complications | 5 year
  Frequency of implant sites with sign of inflammatory reactions with or without marginal bone loss (periimplantitis or peri-implant mucositis). The number of implant sites with bleeding on probing, suppuration or fistula will be registered and described.
Sialometry | 5 year
  measurement of stimulated or unstimulated saliva flow, ml/min for all participants and statistical comparison between the participants in both groups.
Technical outcome | 5 years
  The frequency of prosthetic complications such as fracture or loosening of implant-supported crowns at all implant sites in all participants and comparison between to groups
Aesthetic outcome by Copenhagen Index Scores | 5 year
  Aesthetic parameters:
  Symmetry/harmony, Crown morphology, Crown color match, mucosal discoloration, Papilla Index score mesially and distally Score 1, 2, 3 and 4 (socre 1 for the most optimal and socre 4 for unacceptable aesthetic outcome)
Patient-reported outcome | 5 years
  Oral Health Impact on the Quality of Life (OHIP-49 questionnaire) Response scale from 0 (never experienced problem) to 4 (problem experienced very often).

SECONDARY OUTCOMES:
Decayed, Missing, Filled Tooth index (DMFT) | 5 years
  Caries experience by calculation of total number of tooth with Decayed, Missing or Filled tooth. Less scores indicating better dental condition. Both groups will be compared and the relation to sialometry will be analyzed.
Modified Plaque Index | 5 years
  The Oral hygiene of the patients will be measured by recording the amount of the plaque on the implants and all natural teeth using the following scale:
  (score 1 to 4) Score 1: no visible plaque; Score 2: small amount of hardly visible plaque; Score 3: moderate amount of plaque; Score 4: abundant amount of plaque The difference in plaque index and the relation to the biological complication will be statistically analyzed in both group of participants.
Modified Mucosal Index scores | 5 years
  The sign of inflammatory reactions around the implants will be measured by using the following scores:
  (score 1 to 4) Score 1: normal appearance of gingiva/mucosa; Score 2: slight redness or hyperplasia; Score 3: moderate inflammation with marked redness and hyperplasia and easily bleeding by probing; Score 4: Severe inflammation with severe redness and hyperplasia and spontaneous bleeding The difference in mucosal index and the relation to the plaque index will be statistically analyzed in both group of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Hosseini, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Isidor F, Brondum K, Hansen HJ, Jensen J, Sindet-Pedersen S. Outcome of treatment with implant-retained dental prostheses in patients with Sjogren syndrome. Int J Oral Maxillofac Implants. 1999 Sep-Oct;14(5):736-43. PMID 10531746
- [Result] Pedersen AM, Bardow A, Nauntofte B. Salivary changes and dental caries as potential oral markers of autoimmune salivary gland dysfunction in primary Sjogren's syndrome. BMC Clin Pathol. 2005 Mar 1;5(1):4. doi: 10.1186/1472-6890-5-4. PMID 15740617
- [Result] Hosseini M, Gotfredsen K. A feasible, aesthetic quality evaluation of implant-supported single crowns: an analysis of validity and reliability. Clin Oral Implants Res. 2012 Apr;23(4):453-8. doi: 10.1111/j.1600-0501.2011.02162.x. Epub 2011 Mar 28. PMID 21443589
- [Result] Shiboski SC, Shiboski CH, Criswell L, Baer A, Challacombe S, Lanfranchi H, Schiodt M, Umehara H, Vivino F, Zhao Y, Dong Y, Greenspan D, Heidenreich AM, Helin P, Kirkham B, Kitagawa K, Larkin G, Li M, Lietman T, Lindegaard J, McNamara N, Sack K, Shirlaw P, Sugai S, Vollenweider C, Whitcher J, Wu A, Zhang S, Zhang W, Greenspan J, Daniels T; Sjogren's International Collaborative Clinical Alliance (SICCA) Research Groups. American College of Rheumatology classification criteria for Sjogren's syndrome: a data-driven, expert consensus approach in the Sjogren's International Collaborative Clinical Alliance cohort. Arthritis Care Res (Hoboken). 2012 Apr;64(4):475-87. doi: 10.1002/acr.21591. PMID 22563590